CLINICAL TRIAL: NCT05259943
Title: Microdosing Psychedelics to Improve Mood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rotem Petranker (Other)
Collaborators: Nikean Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Rotem Petranker, Associate Director, Psychedelic Studies Research Program, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ABC123DRM
Record Dates: First submitted 2022-02-15; First posted 2022-03-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: Psilocybin; Psychedelics; Creativity; Mindfulness; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: This trial starts as a placebo-control for 4 weeks and then becomes Open Label for 4 additional weeks. Follow-up assessments will be performed weekly for the first 4 weeks following the last Open Label week.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will not know whether they received placebo or psilocybin in the first stage of the trial.
  Care providers and investigators will not know whether participants received placebo or psilocybin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Blinded Placebo (Placebo Comparator): In this condition participants will receive an inert placebo once weekly for 4 weeks, but they will not know whether they receive placebo or psilocybin.
  Interventions: Drug: Placebo first
- Blinded Psilocybin (Experimental): In this condition participants will receive psilocybin once weekly for 4 weeks, but they will not know whether they receive placebo or psilocybin.
  Interventions: Drug: Psilocybin first
- Open Label (Experimental): In this condition participants will receive psilocybin once weekly for 4 weeks, and will be told that they are receiving psilocybin.
  Interventions: Drug: Psilocybin first; Drug: Placebo first

INTERVENTIONS:
Drug: Psilocybin first — Participants will receive 8 doses of 2mg psilocybin.
  Arms: Blinded Psilocybin; Open Label
Drug: Placebo first — Participants will receive 4 doses of placebo followed by 4 doses of 2mg psilocybin
  Arms: Blinded Placebo; Open Label

SUMMARY:
This trial aims to examine the safety and efficacy of small (2mg) sub-hallucinogenic doses of psilocybin in people with Major Depressive Disorder.

DETAILED DESCRIPTION:
This protocol is for a University of Toronto - sponsored, randomized, placebo-controlled crossover phase 2 study of the safety and efficacy of low doses of psilocybin in subjects with depressive symptoms who meet Diagnostic and Statistical Manual 5 (DSM-5) criteria for diagnosis of a major depressive disorder (MDD) and who are either unwilling to pursue standard treatment (psychotherapy and/or pharmacotherapy) or have previously been non-responsive to standard treatment. This feasibility study will assess whether microdosing has a short-term impact on participant ratings of depressive symptoms. Participants will be administered one dose of either placebo or psilocybin once weekly for four weeks, and then all participants will be administered a dose of psilocybin once weekly for four additional weeks. Short surveys will be collected once weekly three days after the administration of psilocybin/placebo, and follow-ups will occur for up to two years following the beginning of the trial. Using this design will maximize the experimental power to detect an effect if one exists and would inform future research on microdosing in terms of duration, effect size, and expectancy bias.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Have given written informed consent.
* Have a high school level of education.
* Be fluent in speaking and reading the study site's predominantly used or recognized language (i.e., English).
* Be 18 to 65 years old.
* If of childbearing potential, must have a negative pregnancy test at study entry and must agree to use adequate birth control 10 days after the last Experimental Session (refer to section 9.4.2 for contraceptive guidelines).
* Have a preexisting diagnosis of MDD with dysthymic subtype or receive a diagnosis of MDD during screening.
* Agree that for one week preceding each psilocybin session, they will refrain from taking any nonprescription medication, nutritional supplements, or herbal supplement except when approved by the research team. Exceptions will be evaluated by the research team and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals with the exception of SAM-e, 5-HTP, L-tryptophan, and St. John's Wort.
* Agree to consume approximately the same amount of caffeine-containing beverage (i.e. coffee, tea) that they consume on a usual morning, before arriving at the research unit on the mornings of psilocybin session days. Caffeine consumption should not exceed more than ≥600mg/day. If the patient does not routinely consume caffeinated beverages, they must agree not to do so on psilocybin session days.
* Agree not to take any as needed (PRN) medications on the mornings of psilocybin sessions. Non-routine PRN medications for treating breakthrough pain that were taken in the 24 hours before the psilocybin session may result in rescheduling the treatment session, with the decision at the discretion of the investigators.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each psilocybin administration. As described elsewhere, exceptions include daily use of caffeine.

Exclusion Criteria:

* The subject has participated in another investigational study within 60 days prior to the screening visit.
* Cardiovascular conditions: coronary artery disease, uncontrolled hypertension, angina, a clinically significant ECG abnormality (i.e. atrial fibrillation), TIA in the last 6 months, stroke, peripheral or pulmonary vascular disease (no active claudication).
* Blood pressure exceeding screening criteria described below:

  ○ Cardiovascular screening:
  * At the screening and randomization visit, blood pressure will be assessed to qualify to proceed in the trial. Each assessment occasion will involve two or more blood pressure readings. To qualify for the study, the mean blood pressure (mmHg) of the two readings will not exceed 140 systolic and 90 diastolic.
  * Blood pressure (BP) will be taken while subjects are at rest and have been seated or supine for at least 5 minutes. The assessment will involve the average of 2 or more readings separated by fifteen minutes. If the first 2 readings differ by more than 5 mmHg, additional readings will be obtained and averaged. During the BP assessment, the volunteer will be acclimated to the automated blood pressure monitoring equipment by repeatedly taking blood pressure (at least 3 readings) with the device.
* Epilepsy with a history of seizures.
* The subject has a history of cerebral ischemia, transient ischemic attack, intracranial aneurysm, or arteriovenous malformation.
* The subject has a clinically significant history of head injury or head trauma per the judgement of the investigator.
* The subject has a history of cancer.
* Unstable medical condition, severe renal disease (creatinine clearance < 40 ml/min using the Cockcroft and Gault equation), hepatic disease (known history of liver disease, abnormal elevations in LFTs), or serious central nervous system pathology.
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia.
* Are pregnant (positive urine pregnancy test assessed at screening) or nursing, or are of childbearing potential and are not practicing an effective means of birth control (refer to section 9.4.2 for contraceptive guidelines).
* Currently taking on a regular (i.e. daily) basis any psychotropic medications including: investigational agents, psychoactive prescription medications (i.e. benzodiazepines), antidepressants, medications having a primary pharmacological effect on serotonin neurons (i.e. ondansetron), medications that are MAO inhibitors, opioid medications. If previously on antidepressants a minimum of five half lives must have passed from the last dose of medication plus an additional seven days of stabilization before first administration of the drug.
* Current use of any the following of potent metabolic inducers or inhibitors: Inducers - Rifamycin (rifampin, rifabutin, rifapentine), anticonvulsants (carbamazepine, phenytoin, Phenobarbital), Nevirapine, Efavirenz, Taxol, Dexamethasone), St John's Wort; All cytochrome P450 Inhibitors - including all HIV protease inhibitors, verapamil, diltiazem, itraconazole, ketoconazole, erythromycin, clarithromycin, azithromycin, and troleandomycin.
* Use of steroids within the past two weeks.
* Current use of the following drugs will also meet exclusion criteria: ergot alkaloids, pimozide, midazolam, triazolam, lovastatin, simvastatin, fentanyl.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages within 24 hours of each drug administration. The exception is caffeine.
* Must not be a habitual smoker.
* Refrain from starting any new medications.
* Refrain from starting any new complementary or alternative medicine practices (i.e. nutrition/diet modifications, supplements, meditation practice, etc.).
* Are willing to comply with medication requirements per the protocol (refer to Section 6.2).
* Lifestyle Criteria; Refrain from working night shifts.

Psychiatric Exclusion Criteria:

* Current or past history of meeting DSM-V criteria for Schizophrenia, Psychotic Disorder, or Bipolar I or II Disorder.
* Active Major Depressive Disorder Episode.
* Having a first or second-degree relative with schizophrenia, psychotic disorder (unless substance-induced or due to a medical condition), or bipolar I or II disorder.
* Currently meets DSM-V criteria for Dissociative Disorder, Anorexia Nervosa, Bulimia Nervosa, or other psychiatric conditions judged to be incompatible with the establishment of rapport or safe exposure to psilocybin.
* Current or past history within the last 5 years of meeting DSM-V criteria for a moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine).
* Use within 6 months of psychedelic substances.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire Somatic-Anxiety-Depression | Every week until week 4.
  The PHQ-SADS is a 32-item self-report subset of the full PHQ designed to detect the co-occurrence of somatic, anxiety, and depressive symptoms (the SAD triad). Responses are measured using a likert scale between 0 (not bothered) and 2 (bothered a lot). Higher scores suggest more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Psych Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We will pre-register our study and we will make our data available. Whether IPD will be available is TBD.